CLINICAL TRIAL: NCT01677312
Title: Multi-Center Randomized Trial Comparing 19 and 25-gauge Needles for Endoscopic Ultrasound-guided Fine Needle Aspiration (EUS-FNA) of Solid Pancreatic Mass Lesions
Brief Title: Trial Comparing 19 and 25-gauge EUS-FNA Needles
Acronym: EUS-FNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 356077
Record Dates: First submitted 2012-08-28; First posted 2012-09-03 (Estimated); Results first posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Cancer of Pancreas; Pancreatic Neoplasm
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 19G FNA needle (Active Comparator): Evaluate median number of passes to diagnosis (Diagnostic accuracy) and ability to procure histological samples using a 19G FNA needle when performing pancreatic biopsy.
  Interventions: Procedure: Pancreatic Biopsy; Procedure: Histological Samples
- 25G FNA needle (Active Comparator): Evaluate median number of passes to diagnosis (Diagnostic accuracy) and ability to procure histological samples using a 25G FNA needle when performing pancreatic biopsy.
  Interventions: Procedure: Pancreatic Biopsy; Procedure: Histological Samples

INTERVENTIONS:
Procedure: Pancreatic Biopsy — A FNA needle will be used to biopsy the pancreatic mass. The rates of diagnostic accuracy (%) will be assessed. Diagnostic accuracy is defined as the proportion of patients in whom a definitive diagnosis can be obtained within a predetermined number of FNA passes.
Procedure: Histological Samples — The proportion of patients (%) in whom a histological tissue can be obtained when performing a biopsy of the pancreas using a specific needle will be assessed.

SUMMARY:
This study compares the 19G and 25G needles for procuring tissue samples from the pancreas during Endoscopic Ultrasound (EUS) procedures.

DETAILED DESCRIPTION:
The study compares the median number of passes to establish a definitive diagnosis using the 19G or 25G needles. Also, the ability of both needles to procure a histological core tissue is assessed.

ELIGIBILITY:
INCLUSION CRITERIA:

(1) Patients with solid pancreatic mass lesions.

EXCLUSION CRITERIA:

1. Age < 19 years
2. Unable to safely undergo EUS for any reason
3. Coagulopathy (INR > 1.6, Prothrombin Time > 18secs, Thrombocytopenia < 80,000 cells/ml)
4. Unable to consent
5. Non-English speaking patients

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: shyam varadarajulu, MD, Principal Investigator — Florida Hospital Center for Interventional Endoscopy
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Florida Hospital, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- 19G FNA Needle: 19G needle was used for procuring tissue samples from the pancreas during Endoscopic Ultrasound (EUS) procedures
- 25G FNA Needle: 25G needle was used for procuring tissue samples from the pancreas during Endoscopic Ultrasound (EUS) procedures
Period: Overall Study
Arm/Group | 19G FNA Needle | 25G FNA Needle
Started | 36 | 36
Completed | 36 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 19G FNA Needle | 25G FNA Needle | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (9.3) | 67.1 (11.5) | 67.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 21 | 22 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 11 | 18
  White | 28 | 24 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 36 | 36 | 72

OUTCOME MEASURES:

1. Primary Outcome: Median Number of Passes to Establish Diagnosis
Description: To compare the median number of passes required to establish diagnosis using the 19G and 25G needles for FNA of solid pancreatic mass lesions. This will be measured by comparing the rates of diagnostic accuracy (%) between both needle types.
Time Frame: 5 months
Measure: Median (Inter-Quartile Range); unit: No. of passes
Arm/Group | 19G FNA Needle | 25G FNA Needle
Number analyzed (Participants) | 36 | 36
No. of passes | 1 [1 to 1] | 1 [1 to 1]

2. Secondary Outcome: Procurement of Histological Samples
Description: The ability of the 19G and 25G needles to obtain core (histological) tissue will be compared and a significance will be determined.
Time Frame: 30 days
Measure: Number; unit: percentage of participants
Arm/Group | 19G FNA Needle | 25G FNA Needle
Number analyzed (Participants) | 36 | 36
percentage of participants | 86.1 | 33.3

3. Secondary Outcome: Needle Dysfunction
Description: The percentage of cases in which needle dysfunction occurs will be compared between the 19G and 25G needle types. Needle dysfunction will be defined as the need to use more than one FNA needle per lesion in an individual patient.
Time Frame: 2 hours
Measure: Number; unit: percentage of participants
Arm/Group | 19G FNA Needle | 25G FNA Needle
Number analyzed (Participants) | 36 | 36
percentage of participants | 0 | 2.8

4. Secondary Outcome: Complications
Description: The safety profile of the 19 and 25G needles will be compared that includes bleeding, pancreatitis and perforation.
Time Frame: 30 days
Measure: Number; unit: percentage of participants
Arm/Group | 19G FNA Needle | 25G FNA Needle
Number analyzed (Participants) | 36 | 36
percentage of participants | 2.8 | 0

ADVERSE EVENTS:
Time Frame: 10 days
Description: Telephone follow up conducted at 24 hours and 10 days post-procedure
Arm/Group | 19G FNA Needle | 25G FNA Needle
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 1/36 | 0/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 19G FNA Needle (N=36) | 25G FNA Needle (N=36)
Bleeding and fever (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes